# Statistical Analysis Plan (SAP)

Effectiveness of Individualized Dietary
Counseling and Nutritional
Monitoring in Reducing CancerAssociated Cachexia among Female
Breast Cancer Patients: A
Randomized Controlled Trial
07 February, 2024

#### Introduction

This SAP outlines the pre-specified statistical methodology used to evaluate the effectiveness of individualized dietary counseling combined with regular nutritional monitoring in reducing cancer-associated cachexia among female breast cancer patients. The protocol adheres to the CONSORT guidelines.

#### **Objectives**

#### **Primary Objective:**

To assess the effect of individualized dietary counseling and regular nutritional monitoring on cachexia severity using the Mini-CASCO tool after six months.

#### **Secondary Objectives:**

To evaluate changes in:

- Body composition
- Inflammatory and metabolic markers
- Physical performance
- Appetite levels
- Quality of life (QoL)

#### **Study Design**

- **Design:** Prospective, parallel-arm, randomized controlled trial
- Randomization: 1:1 ratio with block-stratified randomization (block size = 4)
- Blinding: Outcome assessors and statisticians were blinded

#### Sample Size Determination

Using G\*Power for repeated-measures ANCOVA:

- Effect size (Cohen's d): 0.5
- Power: 80%Alpha: 0.05
- Estimated N: 64 per group (total 128)
- Final enrollment: 134 randomized; 130 completed (65 per group)

#### **Handling of Missing Data**

Missing data (<5%) addressed via Multiple Imputation (Chained Equations, 10 iterations)</li>

Assumed Missing At Random (MAR)

Sensitivity analyses compared results with and without imputation

#### **Effect Size Estimations**

- Cohen's d: within-group effect size
- Partial eta squared (η²): between-group comparisons
- Interpretation thresholds:
- o d ≥ 0.8 = large
- $\circ$   $\eta^2 \ge 0.14 = large$

#### Software

- Statistical analyses were performed using IBM SPSS Statistics v25.0
- Graphs and tables created using Excel and SPSS

#### **Validation and Sensitivity Analyses**

Key assumptions for ANCOVA validated:

- Normality via Shapiro-Wilk test
- Homogeneity of variance via Levene's test
- Sphericity via Mauchly's test
- Sensitivity analysis excluding imputed data showed similar trends

# **Appendix A: List of Variables**

## **Outcome Measures Table**

| Outcome | Туре | Statistical Test | Covariates | Assumption<br>Checks |
|---|---|---|---|---|
| Change in total Mini-<br>CASCO score | Primary | Repeated-<br>measures<br>ANCOVA | Baseline score | Normality,<br>sphericity<br>(Mauchly's<br>test) |
| Domain-specific Mini-<br>CASCO changes | Secondary | Repeated-<br>measures<br>ANCOVA | Baseline scores | Same as above |
| Within-group differences | Secondary | Paired t-tests | | Normality |
| Between-group effect size | Secondary | Partial eta<br>squared (η²) | | |
| Compliance/adherence | Secondary | Frequency, percentage | | |

## **List of Variables Table**

| Variable | Туре | Tool/Scale |
|-----------------------|-----------------|---------------------------------|
| Weight | Continuous | Digital scale |
| Lean body mass | Continuous | Bioelectrical impedance |
| | | analysis |
| CRP, Albumin, Hb, TLC | Continuous | Blood test |
| ECOG performance | Ordinal | ECOG Scale |
| Appetite | Ordinal | Simplified Nutritional Appetite |
| | | Questionnaire (SNAQ) |
| QoL | Continuous | EORTC QLQ-C30 (Urdu version) |
| Total Mini-CASCO | Composite score | 0–100 scale |